CLINICAL TRIAL: NCT00697333
Title: Optimisation of Radiotherapy-Planning in Patients With Inoperable Locally Advanced Non-Small-Cell Lung Cancer by FDG-PET
Brief Title: Radiotherapy Planning Based on Positron Emission Tomography With Fluoro-deoxyglucose For Advanced NSCLC
Acronym: PET-Plan
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arbeitsgemeinschaft Nuklearmedizin und Strahlentherapie der DEGRO und DGN (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ursula Nestle, Prof. Dr. Ursula Nestle, Universitätsklinikum Freiburg, Arbeitsgemeinschaft Nuklearmedizin und Strahlentherapie der DEGRO und DGN
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG NUK/RT 2006-1
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; FDG-PET; Radiotherapy; planning; target volumes
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (No Intervention): Irradiation of all tumor manifestations detectable by CT and/or positron emission tomography using fluoro-deoxy-glucose including a part of eventual atelectasis and the whole affected lymph node stations by 60 - 74 Gy/2Gy) irradiation of elective lymph node stations up to 50 Gy/2 Gy
- B (Experimental): Irradiation of all tumor manifestations detectable by positron emission tomography using fluoro-deoxy-glucose including the whole affected lymph node stations by 60 - 74 Gy/2Gy
  Interventions: Procedure: restriction of radiotherapy to FDG-PET positive areas only

INTERVENTIONS:
Procedure: restriction of radiotherapy to FDG-PET positive areas only — Restriction of target volumes to areas positive in positron emission tomography using fluoro-deoxy-glucose
  Arms: B

SUMMARY:
Simultaneous radio-chemotherapy in advanced non-small cell lung cancer. The study focusses on a randomised comparison of conventional radiotherapy planning with irradiation of macroscopic tumor and lymph nodes together with prophylactic target volumes vs. irradiation only of FDG-positive lesions.

Primary endpoint is the local disease control in the chest.

DETAILED DESCRIPTION:
Simultaneous radio-chemotherapy in advanced non-small cell lung cancer. The study focusses on a randomised comparison of conventional radiotherapy planning with irradiation of macroscopic tumor and lymph nodes together with prophylactic target volumes vs. irradiation only of FDG-positive lesions.

Primary endpoint is the local disease control in the chest

ELIGIBILITY:
Inclusion Criteria:

* histologically proved NSCLC
* UICC-stage I-III, no resection planned
* complete staging < 6 wks before treatment including cranial CT
* ECOG <3, Karnofsky-Index >60%
* age > 18 <
* FEV1 > 1,0 l or >35%
* RT-planning according to protocol feasible
* chemotherapy feasible
* written informed consent

Exclusion Criteria:

* neuroendocrine tumors, plain broncho-alveolar-cell ca.
* distant metastases, supraclavicular lymph node metastases
* malignant pleural effusion
* resection of actual tumor performed
* inclusion in other study protocol
* chemotherapy due to actual tumor before FDG-PET
* induction-chemotherapy
* acute vena cava superior syndrome
* second malignancy other than basalioma
* pregnancy, lactation
* heart insufficiency NYHA III/IV
* pneumoconiosis with active inflammatory changes of mediastinal lymph nodes
* acute broncho-pulmonary infection at time of PET-examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-05; Primary Completion 2016-11 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
time to local progression | actuarial
  Time from randomization to first evidence of local progression or last follow up

SECONDARY OUTCOMES:
Overall survival | actuarial
  Time from randomization to death or last follow up
normal tissue toxicity | actuarial
  Time from randomization to death or last follow up
in and out field progression | actuarial
  Time from randomization to progression or last follow up

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Nestle, Prof., Principal Investigator — Universitätsklinikum Freiburg, Germany
Locations (2):
- Germany (2):
  - Universitätsklinikum Freiburg, Freiburg I. Br., Baden-Wurttemberg
  - Universitätsklinikum Freiburg, Freiburg i.Br., Baden-Wurttemberg

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Nestle U, Kremp S, Grosu AL. Practical integration of [18F]-FDG-PET and PET-CT in the planning of radiotherapy for non-small cell lung cancer (NSCLC): the technical basis, ICRU-target volumes, problems, perspectives. Radiother Oncol. 2006 Nov;81(2):209-25. doi: 10.1016/j.radonc.2006.09.011. Epub 2006 Oct 24. PMID 17064802
- [Background] Nestle U, Schaefer-Schuler A, Kremp S, Groeschel A, Hellwig D, Rube C, Kirsch CM. Target volume definition for 18F-FDG PET-positive lymph nodes in radiotherapy of patients with non-small cell lung cancer. Eur J Nucl Med Mol Imaging. 2007 Apr;34(4):453-62. doi: 10.1007/s00259-006-0252-x. Epub 2006 Oct 21. PMID 17058078
- [Background] Nestle U, Kremp S, Schaefer-Schuler A, Sebastian-Welsch C, Hellwig D, Rube C, Kirsch CM. Comparison of different methods for delineation of 18F-FDG PET-positive tissue for target volume definition in radiotherapy of patients with non-Small cell lung cancer. J Nucl Med. 2005 Aug;46(8):1342-8. PMID 16085592
- [Background] MacManus M, Nestle U, Rosenzweig KE, Carrio I, Messa C, Belohlavek O, Danna M, Inoue T, Deniaud-Alexandre E, Schipani S, Watanabe N, Dondi M, Jeremic B. Use of PET and PET/CT for radiation therapy planning: IAEA expert report 2006-2007. Radiother Oncol. 2009 Apr;91(1):85-94. doi: 10.1016/j.radonc.2008.11.008. Epub 2008 Dec 25. PMID 19100641
- [Background] Nestle U, Weber W, Hentschel M, Grosu AL. Biological imaging in radiation therapy: role of positron emission tomography. Phys Med Biol. 2009 Jan 7;54(1):R1-25. doi: 10.1088/0031-9155/54/1/R01. Epub 2008 Dec 5. PMID 19060363
- [Background] Schaefer A, Kremp S, Hellwig D, Rube C, Kirsch CM, Nestle U. A contrast-oriented algorithm for FDG-PET-based delineation of tumour volumes for the radiotherapy of lung cancer: derivation from phantom measurements and validation in patient data. Eur J Nucl Med Mol Imaging. 2008 Nov;35(11):1989-99. doi: 10.1007/s00259-008-0875-1. Epub 2008 Jul 26. PMID 18661128
- [Derived] Craddock M, Nestle U, Koenig J, Schimek-Jasch T, Kremp S, Lenz S, Banfill K, Davey A, Price G, Salem A, Faivre-Finn C, van Herk M, McWilliam A. Cardiac Function Modifies the Impact of Heart Base Dose on Survival: A Voxel-Wise Analysis of Patients With Lung Cancer From the PET-Plan Trial. J Thorac Oncol. 2023 Jan;18(1):57-66. doi: 10.1016/j.jtho.2022.09.004. Epub 2022 Sep 18. PMID 36130693
- [Derived] Nestle U, Schimek-Jasch T, Kremp S, Schaefer-Schuler A, Mix M, Kusters A, Tosch M, Hehr T, Eschmann SM, Bultel YP, Hass P, Fleckenstein J, Thieme A, Stockinger M, Dieckmann K, Miederer M, Holl G, Rischke HC, Gkika E, Adebahr S, Konig J, Grosu AL; PET-Plan study group. Imaging-based target volume reduction in chemoradiotherapy for locally advanced non-small-cell lung cancer (PET-Plan): a multicentre, open-label, randomised, controlled trial. Lancet Oncol. 2020 Apr;21(4):581-592. doi: 10.1016/S1470-2045(20)30013-9. Epub 2020 Mar 12. PMID 32171429
- [Derived] Nestle U, Rischke HC, Eschmann SM, Holl G, Tosch M, Miederer M, Plotkin M, Essler M, Puskas C, Schimek-Jasch T, Duncker-Rohr V, Ruhl F, Leifert A, Mix M, Grosu AL, Konig J, Vach W. Improved inter-observer agreement of an expert review panel in an oncology treatment trial--Insights from a structured interventional process. Eur J Cancer. 2015 Nov;51(17):2525-33. doi: 10.1016/j.ejca.2015.07.036. Epub 2015 Aug 12. PMID 26277100